CLINICAL TRIAL: NCT05112653
Title: Value of MicroRNA30a in Philadelphia Positive Leukemic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager mohammed, assuit university, Assiut University
Other Study IDs: AssiutU2021
Record Dates: First submitted 2021-07-10; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Possibility of Using microRNA30a as a Prognostic Marker in Philadelphia Positive Leukemic Patients by Measure Level of microRNA30a in Blood Sample

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 2: Group of Philadelphia positive leukemic patients will included in the study who divide into:
  * patient newly diagnosed CML treated with first line of tyrosine kinase inhibitors therapy.
  * Philadelphia positive acute leukemic patients(ALL, mixed-phenotype acute leukemia) on TKI therapy who achieved complete hematological remission(CHR) and who failed to achieve CHR.

SUMMARY:
The Philadelphia chromosome in leukemogenesis:The truncated chromosome 22 that results from the reciprocal translocation t(9;22)(q34;q11) is known as (Ph) and is a hallmark of (CML). This aberrant fusion gene encodes the breakpoint cluster region-proto-(BCR-ABL1) oncogenic protein with persistently enhanced tyrosine kinase activity. Besides CML, the Ph is found in acute lymphoblastic leukemia, and mixed-phenotype acute leukemia.

Chronic myeloid leukemia is a myeloproliferative neoplasm, characterized by the unrestrained expansion of pluripotent bone marrow stem cells.The hallmark of the disease is the presence of a reciprocal t(9;22)(q34;q11.2), resulting in a derivative 9q+ and a small 22q-. The latter, known as the Philadelphia chromosome, results in a BCR-ABL fusion gene . The diagnosis requires fluorescent in situ hybridization (to demonstrate the BCR-ABL fusion gene or(PCR) to demonstrate the BCR-ABL mRNA transcript.

DETAILED DESCRIPTION:
our study will discuss the possible value of microRNA30a as early predictor for TKIs resistance in newly diagnosed CML patients.

the study will dectect the possible value of microRNA30a as prognostic marker in Philadelphia positive acute leukemic patients(ALL, mixed-phenotype acute leukemia) on TKI therapy by assessment level of microRNA30a inpatients who achieved complete hematological remission(CHR) and who failed to achieve CHR.

The study goal has been taken through the role of microRNA30a in reducing ABL1 and BCR-ABL1 protein expression and microRNAs are capable of changing the levels of several key proteins at various steps of the autophagic pathway.

ELIGIBILITY:
3 a-Inclusion criteria

1_clinical diagnosis of Philadelphia positive leukemic patients (males and females).

2- Aged from 18- 60 years. 3-All eligible patients presenting at Clinical Haematology Unit Internal Medicine Department.

4- Without contraindication to receive TKIs therapy. 5-Must able to swallow tablet(TKI therapy).

-exclusion criteria

1. NO bone marrow aspirate and flow cytometry confirm their diagnosis.
2. patients who refuse to participate in the study.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Gender Based: Yes — more in males
Study Population: 70 patients diagnosed as Philadelphia positive leukemic patients(CML, acute lymphoblastic leukemia, and mixed-phenotype acute leukemia).
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To detect the possibility of using microRNA30a as a prognostic marker in Philadelphia Positive Leukemic Patients by measure level of microRNA30a in blood sample of Philadelphia positive leukemic patients on tyrosine kinase inhibitor therapy | 2 years
  The study goal has been taken through the role of microRNA30a in reducing ABL1 and BCR-ABL1 protein expression and microRNAs are capable of changing the levels of several key proteins at various steps of the autophagic pathway.